CLINICAL TRIAL: NCT03881085
Title: The Science of Behavior Change in African American Breast Cancer Survivors
Brief Title: Stress Reactivity Among African American Breast Cancer Survivors
Status: Completed | Type: Observational
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Sponsor
Other Study IDs: AABCSR
Record Dates: First submitted 2019-03-04; First posted 2019-03-19 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Breast Cancer Female; Stress Reaction
Keywords: minorities; stress reactivity; allostatic load; disparities
MeSH Terms: conditions — Fractures, Stress

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples, urine samples, and saliva samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Despite increased access to early detection and the availability of more effective therapeutic strategies, African American women continue to experience excess rates of morbidity and mortality from breast cancer. An emerging hypothesis about breast cancer disparities is that social conditions and physiological responses to social stressors influence biological processes that are important to the initiation and progression of disease. This hypothesis is based on data from animal studies which have shown that rats that are exposed to social stressors such as isolation are likely to develop mammary tumors that are histologically and etiologically similar to those that develop among African American women. The HPA axis plays a central role in regulating the physiological stress response; dysregulation of the HPA has been suggested as a mechanism through which social and biological factors contribute to racial disparities in breast cancer outcomes. Many African Americans experience stressful life events and circumstances, including economic, discriminatory, and other stressors. These social factors may contribute to an increased risk of advanced stage disease, but not all African American women who are exposed to adverse social factors develop advanced stage disease and those who have a limited number of psychosocial stressors can develop advanced stage breast cancer, regardless of early detection. This may be because stress reactivity, or one's physiological and psychological responses to a stressor, is highly individualized and dependent on psychological and social determinants as well as genetic factors. But, these biological and psychosocial pathways have not been examined among women at increased risk for disparities. Therefore, this study will characterize stress reactivity and emotional regulation among African American breast cancer survivors and measure the association between these responses and decisions about cancer control and treatment compliance. As part of providing empirical data on biological and psychological pathways that contribute to breast cancer disparities, the investigator's study will identify novel intervention targets that can be used to improve self-management in a population that is at risk for limited cancer control.

DETAILED DESCRIPTION:
Dysregulation of the HPA has been suggested as a mechanism through which social and biological factors contribute to racial disparities in breast cancer outcomes.The HPA axis plays a central role in regulating the physiological stress response;a prolonged and elevated glucocorticoid (GC) response following a social stressor predicts tumor growth rates and the development of mammary cancer in rats that histologically and etiologically resembles human disease.Many African Americans experience stressful life events and circumstances, including economic, discriminatory, and other stressors. These psychosocial factors may contribute to an increased risk of advanced stage breast cancer among African American women, but not all African American women who are exposed to adverse psychosocial and social stressors develop advanced stage breast cancer and African American women who have a limited number of stressors also develop advanced stage breast cancer, regardless of early detection. This may be because stress reactivity, or one's physiological and psychological responses to a stressor, is highly individualized and dependent on psychological and social determinants. However, empirical data are not available on stress reactivity among African American breast cancer survivors and how these reactions vary among women based on their exposure to chronic stressors and psychological characteristics. Empirical data are also lacking on the association between stress reactivity and cancer control behaviors among African American breast cancer survivors even though prior studies have shown that these women are less likely than whites to engage in health behaviors that are important to cancer control and research is now being conducted to understand how stress affects these behaviors.This research is testing the hypothesis that stress: (1) promotes temporal discounting; (2) has an adverse effect on self-efficacy, and (3) reduces executive functioning (e.g., goal setting, planning). However, stress reactivity, and the association between these responses and cancer control behaviors (e.g., diet, physical activity, and treatment compliance), have not been examined among African American breast cancer survivors. Prior studies have shown that African Americans have a dysregulated stress response as a result of persistent exposure to chronic and acute and stressors; this may alter stress responses and lead to high levels of allostatic load. In order to develop effective behavioral interventions for African American breast cancer survivors, an important first step is to verify that the mechanisms (e.g., temporal discounting, self-efficacy) involved in health behaviors for cancer control (e.g., diet, physical activity, treatment compliance) are associated with stress reactivity among these women. Therefore this study will characterize stress reactivity among African American breast cancer survivors and validate the association between these responses and targeted mechanisms of behavior change.

ELIGIBILITY:
Inclusion Criteria:

* Self-identify as African American or Black women
* Histologically confirmed stage of I, II, or IIIa breast cancer.
* Between the ages of 21-75 at diagnosis
* Have been diagnosed within the last 5 years

Exclusion Criteria:

* Women who are not African American or Black
* Diagnosed with a later stage of breast cancer
* Not within the defined treatment parameters

Ages: 21 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Due to the nature of this study, only women who were born biologically as female will be eligible to participate in this study. Men who develop breast cancer have a different pathophysiology than women, and therefore, will not be included in this sample.
Study Population: Subjects eligible to participate in this study include African American breast cancer survivors who were diagnosed with Stage I, II, or Illa disease and have completed all breast cancer treatment. Women who are both acute and long-term survivors are eligible to participate in this study. For all women, patients must have been between the ages of 21-75 at diagnosis and diagnosed within the last 5 years. For those who are acute survivors, patients are eligible to participate in the study if they completed surgical treatment within the past three months, regardless of if they have initiated adjuvant therapy.
Sampling Method: Non-Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2018-10-19 (Actual); Primary Completion 2021-07-20 (Actual); Study Completion 2021-07-20 (Actual)

PRIMARY OUTCOMES:
Examine stress reactivity among African American Breast Cancer Survivors utilizing cortisol. | 21 months
  Conduct an A Tier Social Stress Test (TSST)with patients to induce a stress response. Cortisol is being examined as a stress biomarker and will be measured at baseline, at multiple timepoints (n=3) during the TSST, and immediately after the TSST to assess changes in cortisol levels.
Examine stress reactivity among African American Breast Cancer Survivors utilizing vital signs. | 21 months
  Collect vital assessments that include heart rate and systolic and diastolic blood pressure at baseline, during the course of the Trier Social Stress Test (TSST), and immediately after the TSST in order to examine changes in vitals as it relates to stress responses during the TSST.
Examine the association between levels of stress reactivity and stressors as it relates to socioeconomic status, clinical factors, and social stress | 21 months
  Characterize the nature and distribution of stress reactivity among African American breast cancer survivors based on socioeconomic, clinical, and social stressors. Socioeconomic status will be collected via self-report utilizing household income and education items from the Behavioral Risk Factor Surveillance System (BRFSS) tool. Financial strain will be evaluated using the Comprehensive Score for financial Toxicity (COST) tool. Social stress will be assessed by levels of social isolation using the loneliness scale. Clinical variables relating to disease stage will be extracted from the patient's electronic medical record.
Examine glucocorticoid sensitivity as a potential predictor of stress reactivity | 21 months
  A blood sample will determine circulating levels of neutrophils, lymphocytes, and monocytes to determine glucocorticoid sensitivity.
Examine stress reactivity on temporal discounting | 21 months
  The Kirby Delay Discounting Task conducted immediately (10 minutes) or longer (20 minutes) following exposure to the Trier Social Stress Test to examine temporal discounting.
Determine the extent to which active engagement with a stressor is associated with adherence to dietary recommendations for cancer control | 1 month
  Self-reported diet behaviors will be associated with levels of stress reactivity 1-month following stress induction.
Determine the extent to which active engagement with a stressor is associated with adherence to physical activity recommendations for cancer control | 1 month
  Self-reported physical activity behaviors will be associated with levels of stress reactivity 1-month following stress induction.

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Halbert CH, Jefferson MS, Danielson C, Froeliger B, Giordano A, Thaxton JE. An observational study and randomized trial of stress reactivity in cancer disparities. Health Psychol. 2020 Sep;39(9):745-757. doi: 10.1037/hea0000882. PMID 32833476